CLINICAL TRIAL: NCT01649180
Title: NEXT: Subsequent Exposure to Tyrosine Kinase Inhibition (TKI) at Recurrence After Adjuvant Therapy in Renal Cell Carcinoma (RCC)
Brief Title: NEXT: Subsequent Exposure to Tyrosine Kinase Inhibition at Recurrence After Adjuvant Therapy in Renal Cell Carcinoma
Acronym: PrE0801
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to prolonged enrollment timelines
Sponsor: PrECOG, LLC. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PrE0801; WS1512227 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2012-07-21; First posted 2012-07-25 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; Clear Cell Renal Cell Carcinoma; ccRCC; Metastatic RCC; Recurrent RCC; Kidney Cancer; Kidney Neoplasms; Axitinib; AG-013736; Tyrosine Kinase Inhibition; TKI
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Axitinib; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (Experimental): Axitinib will be given orally and will continue until progression of disease.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib 5 mg orally with food every 12 hours. One cycle=28 days.
  Other Names: AG-013736; Tyrosine Kinase Inhibitor (TKI)

SUMMARY:
The purpose of this study is to see how well the study drug, axitinib, helps control renal (kidney) cancer that has come back (recurrent) or spread (metastatic). Patients must have already been treated as a participant in a clinical trial with sunitinib, sorafenib, pazopanib or placebo (sugar pill) after their initial surgery.

This study will examine the effect of adjuvant tyrosine kinase inhibition (TKI) therapy (sorafenib, sunitinib or pazopanib) on subsequent exposure to TKI with axitinib in the first-line recurrent or metastatic setting.

DETAILED DESCRIPTION:
Approximately 64,770 cases of cancer involving the kidney and renal pelvis were diagnosed in the United States in 2012 and 13,570 deaths occurred from these tumors. The rate of Renal Cell Carcinoma (RCC) has increased by 2% per year for the past 65 years. The reason for this increase in unknown but smoking and obesity are risk factors for the development of RCC. Early stage disease is typically treated with resection with definitive intent with partial or radical nephrectomy. Patients with metastatic disease are often treated with systemic therapy with palliative intent. Systemic therapeutic options include so-called targeted therapies, and less often chemotherapy and immunomodulatory therapies (interferon alpha and interleukin-2).

The Food and Drug Administration (FDA) has approved six targeted agents for the treatment of advanced and metastatic renal cell carcinoma that fall into two general classes - vascular endothelial growth factor (VEGF) inhibitors and inhibitors of mammalian target of rapamycin (mTOR). On the basis of several randomized phase III studies, vascular endothelial growth factor receptor-2 (VEGFR2) inhibitor therapy has become the generally preferred treatment for recurrent and metastatic ccRCC (clear cell Renal Cell Carcinoma) in the first-line setting. Treatment of ccRCC with VEGF-inhibition in the first-line metastatic setting, is associated with a progression-free survival of approximately 11 months. Vascular endothelial growth factor (VEGF) inhibitor therapy in the second-line remains active, but to a lesser degree - progression-free survival (PFS) has been reported to be between 5 and 7 months.

Adjuvant treatment of high-risk, early-stage ccRCC with VEGFR2 TKI therapy following definitive resection has become an area of active investigation. The ASSURE trial (ECOG 2805) recently completed accrual, and other adjuvant trials - i.) SORCE (sorafenib for 3 or 1 year versus placebo), ii.) S-Trac (sunitinib versus placebo) - are in accrual.

Axitinib (AG-013736, Pfizer Inc.), a receptor-tyrosine kinase inhibitor that is selective for VEGFR1, 2, and 3, is an important new agent for use in metastatic RCC. Axitinib has been examined extensively in RCC, and it has been shown to be safe, well-tolerated, and highly active. On January 27, 2012, the FDA approved axitinib for the treatment of advanced RCC after failure of one prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent or metastatic RCC requiring systemic therapy following treatment (tx) with sorafenib, sunitinib, pazopanib, or placebo on an adjuvant study
* Required to have primary or recurrence tumor samples containing clear cell variant RCC with <50% of any other histology
* Recurrence must occur ≥ 3 months following end of exposure to the adjuvant intervention
* Received ≥ 3 six week cycles of prior adjuvant tx with sorafenib, sunitinib, pazopanib or placebo in the adjuvant setting on a clinical trial, or recurrence >3 months of tx on an adjuvant placebo arm
* Required to have measurable recurrent or metastatic disease that is not curable by standard radiation therapy or surgery
* Male or female, ≥ 18 years old
* ECOG PS 0 or 1
* Blood pressure (B/P) must be controlled at time of enrollment. Tx with antihypertensive medication(s) is allowed. Controlled B/P is defined as in clinic measurement of systolic B/P ≤ 140 mm Hg AND diastolic B/P ≤ 90 mm Hg. If B/P is uncontrolled at time of planned enrollment, tx or optimization with antihypertensive medication(s) may be initiated in order to control B/P. Patient may be considered for enrollment when this has happened.
* Women must not be pregnant or breastfeeding
* Men and women who are of reproductive potential must be willing to employ an effective method of birth control/contraception
* Willingness and ability to comply with scheduled visits, tx plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign an IRB-approved informed consent
* Adequate organ function as evidenced by the following, obtained within 28 days prior to registration:

  * Absolute neutrophil count (ANC) ≥ 1250 cells/mm³
  * Platelet count ≥ 75,000 cells/mm³
  * Hemoglobin ≥ 9.0 g/dL
  * Total direct serum bilirubin ≤ 1.5x upper limit of normal (ULN)
  * ALT and AST ≤ 2.5 x ULN unless there are liver metastases in which case AST and ALT ≤ 5.0 x ULN
  * Serum creatinine <1.5 x ULN or calculated creatinine clearance ≥ 45 mL/min
  * Urine protein <2+ by urine dipstick
* Resolution of all previous tx-related toxicity to ≤ grade 1 or back to baseline
* No major surgery <4 weeks or radiation therapy <2 weeks of starting study tx. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* No clinically significant gastrointestinal abnormalities
* No current use or anticipated need for tx with drugs that are known potent CYP3A4 inhibitors
* No current or anticipated need for tx with drugs that are known CYP3A4 or CYP1A2 inducers
* No current requirement of anticoagulant therapy with oral vitamin K antagonists
* No untreated brain metastases, spinal cord compression, or carcinomatous meningitis. Patients must be off oral (systemic) steroids prior to registration. Inhalational steroids, e.g., for asthma, emphysema are permissible.
* No serious uncontrolled medical disorder or active infection that would impair their ability to receive study tx
* None of the following conditions within the 6 months prior to study drug: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis or pulmonary embolism
* No known HIV or AIDS-related illness
* No other active malignancy
* No dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol
* No other severe acute/chronic medical or psychiatric condition or lab abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Keefe, MD, Study Chair — University of Pennsylvania Health System
Locations (3):
- United States (3):
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Background] Rini BI, Wilding G, Hudes G, Stadler WM, Kim S, Tarazi J, Rosbrook B, Trask PC, Wood L, Dutcher JP. Phase II study of axitinib in sorafenib-refractory metastatic renal cell carcinoma. J Clin Oncol. 2009 Sep 20;27(27):4462-8. doi: 10.1200/JCO.2008.21.7034. Epub 2009 Aug 3. PMID 19652060
- [Background] Hu-Lowe DD, Zou HY, Grazzini ML, Hallin ME, Wickman GR, Amundson K, Chen JH, Rewolinski DA, Yamazaki S, Wu EY, McTigue MA, Murray BW, Kania RS, O'Connor P, Shalinsky DR, Bender SL. Nonclinical antiangiogenesis and antitumor activities of axitinib (AG-013736), an oral, potent, and selective inhibitor of vascular endothelial growth factor receptor tyrosine kinases 1, 2, 3. Clin Cancer Res. 2008 Nov 15;14(22):7272-83. doi: 10.1158/1078-0432.CCR-08-0652. PMID 19010843
- [Background] Rixe O, Bukowski RM, Michaelson MD, Wilding G, Hudes GR, Bolte O, Motzer RJ, Bycott P, Liau KF, Freddo J, Trask PC, Kim S, Rini BI. Axitinib treatment in patients with cytokine-refractory metastatic renal-cell cancer: a phase II study. Lancet Oncol. 2007 Nov;8(11):975-84. doi: 10.1016/S1470-2045(07)70285-1. Epub 2007 Oct 23. PMID 17959415
- [Background] Escudier B, Gore M. Axitinib for the management of metastatic renal cell carcinoma. Drugs R D. 2011;11(2):113-26. doi: 10.2165/11591240-000000000-00000. PMID 21679004

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axitinib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 54 [52 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to disease progression or death, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessed every 12 weeks up to 36 months
Population: all participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 3
months | 16.6 [16.6 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Secondary Outcome: Overall Response Rate
Description: Best overall response was evaluated using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v 1.0). Response is defined as complete response or partial response.
  Complete Response (CR): disappearance of all target lesions Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Assessed every 12 weeks up to 36 months
Population: all participants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 3
proportion of participants | 1.00 [0.29 to 1.00]

3. Secondary Outcome: Biospecimen Banking for IL-8 and VEGF-A
Description: To bank biospecimens for the retrospective determination of whether baseline or changes in cytokine levels of IL-8 and VEGF-A predict response to treatment in this setting. Banking of plasma and serum is optional but strongly encouraged.
  Note: The assays to assess cytokine levels of IL-8 and VEGF-A were not performed because the study stopped early and only 3 patients were enrolled. Therefore, the analysis to evaluate the associations between response and IL-8 as well as VEGF-A was not done.
Time Frame: Baseline and 8 weeks
Population: Only 3 patients were enrolled. Analysis to evaluate the associations between response and IL-8 as well as VEGF-A was not done.
Arm/Group | Axitinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Biospecimen Banking for SNPs Analysis
Description: To bank biospecimens for the retrospective determination of whether baseline single nucleotide polymorphisms (SNPs) in angiogenesis-related genes predict response to treatment (candidate gene approach). Banking of PBMC is optional but strongly encouraged.
  Note: The SNP genotyping analysis was not performed because the study stopped early and only 3 patients were enrolled. Therefore, the analysis to evaluate the association between baseline SNPs in angiogenesis-related genes and response was not be done.
Time Frame: Baseline
Population: Only 3 patients were enrolled. Analysis to evaluate the association between baseline SNPs in angiogenesis-related genes and response was not be done.
Arm/Group | Axitinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Tumor Tissue Banking
Description: To bank tumor tissue (formalin-fixed, paraffin-embedded tumor blocks) for retrospective examination of the molecular pathophysiologic mediators of tumorigenesis and progression such as phospho-protein expression of MAPK signaling network intermediates in endothelial cells. Banking of tumor tissue is optional but strongly encouraged.
  Note: None of the 3 patients submitted tumor tissues so the analysis won't be performed.
Time Frame: Baseline
Population: None of the 3 patients submitted tumor tissues so the analysis was unable to be performed.
Arm/Group | Axitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed while on treatment (up to 26 months) and for 30 days after the last dose of study drug.
Description: Adverse events were routinely assessed by the treating clinician according to the schedule above.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=3)
Retinal vascular disorder (Eye disorders) | 1 (1) — retinal vein occlusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=3)
Hypertension (Vascular disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No